CLINICAL TRIAL: NCT06539507
Title: A Phase 1/1b Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Single and Multiple Ascending Doses of BCX17725 in Healthy Participants and Multiple Doses of BCX17725 in Participants With Netherton Syndrome
Brief Title: A Study of the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of BCX17725
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: BCX17725-101; U1111-1303-9510 (Other: WHO UTN); 2025-521973-16 (EudraCT Number)
Record Dates: First submitted 2024-07-30; First posted 2024-08-06 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Netherton Syndrome
Keywords: First-in-human; Single ascending dose; Multiple ascending dose; Pharmacokinetics; Placebo control; Netherton syndrome
MeSH Terms: conditions — Netherton Syndrome

STUDY DESIGN:
Intervention Model Description: In Parts 1 and 2, participants will be randomized to BCX17725 or placebo under double-blind conditions. In Parts 3 and 4, participants will receive open-label BCX17725.
Who Masked: Participant, Investigator
Masking Description: Parts 1 and 2 will be blinded; Parts 3 and 4 will be open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Part 1 - BCX17725 single dose (Experimental): Participants randomized to BCX17725 will receive BCX17725 as a single dose in sequential ascending dose cohorts
  Interventions: Drug: BCX17725
- Part 1 - placebo single dose (Experimental): Participants randomized to placebo will receive placebo as a single dose
  Interventions: Drug: Placebo
- Part 2 - BCX17725 multiple doses (Experimental): Participants randomized to BCX17725 will receive BCX17725 as multiple doses in sequential ascending dose cohorts
  Interventions: Drug: BCX17725
- Part 2 - placebo multiple doses (Experimental): Participants randomized to placebo will receive placebo as multiple doses
  Interventions: Drug: Placebo
- Part 3 - BCX17725 multiple doses (Experimental): Participants will receive BCX17725 as multiple doses
  Interventions: Drug: BCX17725
- Part 4 - BCX17725 multiple doses (Experimental): Participants will receive BCX17725 as multiple doses
  Interventions: Drug: BCX17725

INTERVENTIONS:
Drug: BCX17725 — BCX17725 for injection
  Arms: Part 1 - BCX17725 single dose; Part 2 - BCX17725 multiple doses; Part 3 - BCX17725 multiple doses; Part 4 - BCX17725 multiple doses
Drug: Placebo — Placebo for injection
  Arms: Part 1 - placebo single dose; Part 2 - placebo multiple doses

SUMMARY:
This is a first-in-human, Phase 1/1b, 4-part study that includes the evaluation of safety, tolerability, pharmacokinetics (PK), and immunogenicity of BCX17725 when administered via single and multiple doses in healthy adult participants (Parts 1 and 2), and multiple doses in adult participants with Netherton syndrome (Part 3). In Part 4, the effectiveness, safety, and tolerability of BCX17725 when administered via multiple IV and/or SC doses through 12 weeks will be evaluated in adult and adolescent participants with Netherton syndrome.

DETAILED DESCRIPTION:
Parts 1 and 2 are randomized, placebo-controlled, single-ascending-dose (SAD) and multiple-ascending-dose (MAD) study parts, respectively, in healthy participants. Part 3 will evaluate multiple dose administrations in participants with Netherton syndrome in an open-label design. Part 4 will evaluate multiple administrations of BCX17725 in participants with Netherton syndrome in an open-label study design over 12 weeks, with an 8-week post-treatment follow-up period.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or non-pregnant, non-lactating female aged 18 to 55 years, inclusive (Parts 1 and 2), 18 to 65 years, inclusive (Part 3), or 12 to 65 years, inclusive (Part 4)
* Confirmed diagnosis of Netherton syndrome (Parts 3 and 4)
* IGA score of ≥ 3 (Parts 3 and 4) and IASI score of ≥ 16 (Part 4)
* BMI between 18 and 30 kg/m^2, inclusive (Parts 1 and 2)
* Estimated glomerular filtration rate (eGFR) of ≥ 90 mL/min/1.73 m^2 (Parts 1 and 2) or ≥ 60 mL/min/1.73 m^2 (Part 3)
* Agree to follow the protocol contraception requirements from screening until 90 days after the last dose of study drug
* In the opinion of the investigator, expected to adequately comply with all required study procedures and restrictions for the duration of the study

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | From screening through EOS (ie, through Day 78 in Parts 1 and 3, and Day 106 in Part 2)
  Incidence of TEAEs as assessed by Common Terminology Criteria for Adverse Events (CTCAE) from screening through end-of-study (EOS) in each study part
Change from baseline in Ichthyosis Area and Severity Index (IASI) score at Week 12 (Part 4) | From baseline to Week 12
  IASI measures the severity of erythema (IASI-E) and scaling (IASI-S); the maximum sub-scores for the IASI-E and IASI-S being 24, and the maximum total IASI score being 48. Higher scores indicate worse clinical outcome.

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) | Up to Day 64 (Part 1), Day 92 (Part 2), and Day 78 (Part 3)
  Cmax of BCX17725
Time to maximum observed serum concentration (Tmax) | Up to Day 64 (Part 1), Day 92 (Part 2), and Day 78 (Part 3)
  Time to Cmax of BCX17725
Area under the serum concentration-time curve (AUC) from time 0 to the time of last measurable concentration (AUC0-t) | Up to Day 64 (Part 1), Day 92 (Part 2), and Day 78 (Part 3)
  AUC0-t of BCX17725
Terminal elimination half-life (t1/2) | Up to Day 64 (Part 1), Day 92 (Part 2), and Day 78 (Part 3)
  Terminal elimination half-life (t1/2) of BCX17725
Number of participants who are anti-drug antibody (ADA)-positive (baseline and post-baseline) and number of participants who have treatment-emergent ADAs | Day 1 pre-dose and up to Day 64 (Part 1), Day 92 (Part 2), and Day 78 (Part 3)
  Incidence of ADAs to BCX17725
Change from baseline in Investigator Global Assessment (IGA) score at Week 12 (Part 4) | From baseline to Week 12
  IGA assesses the overall severity of a participant's NS skin disease based on a 5-point scale (0, clear; 1, almost clear; 2, mild; 3, moderate; and 4, severe). Higher scores indicate worse clinical outcome.
Change from baseline in Worst Itch Numerical Rating Score (NRS) at Week 12 (Part 4) | From baseline to Week 12
  Worst Itch Numerical Rating Scale (NRS) is a self-rated, single-item scale designed for assessing the worst itch in the past 7 days. The scale uses an 11-point NRS, scored from 0 (no itch) to 10 (worst possible itch). Higher scores indicate worse clinical outcome.
Incidence of TEAEs (Part 4) | From baseline through Week 20
  Incidence of TEAEs as assessed by CTCAE
Serum concentrations of BCX17725 (Part 4) | From baseline through Week 20
  Serum concentrations of BCX17725

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Investigative site, New Haven, Connecticut
  - Investigative site, Indianapolis, Indiana
- Australia (2):
  - Investigative site, Sydney, New South Wales
  - Investigative site, Brisbane, Queensland

IPD SHARING:
Plan to Share IPD: No